CLINICAL TRIAL: NCT05497960
Title: Evaluating the Feasibility and Acceptability of Vivo, an Online, Live and Interactive Strength Training Program, in Sedentary Older Adults With Prediabetes.
Brief Title: Vivo Prediabetes Study: Online, Live, and Interactive Strength Training for Older Adults With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Levian (Industry)
Collaborators: Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Eric Levian, CEO, Impactiv, Inc.
Organization: Impactiv, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00110021; 1R44AG076087-01 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: PreDiabetes; Older Adults; Muscle Loss; Muscle Weakness
Keywords: older adults; pre diabetes; strength training; muscle weakness; resistance training; virtual; intervention
MeSH Terms: conditions — Prediabetic State; Muscular Atrophy; Muscle Weakness; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vivo strength training (Other): Participants will exercise virtually, 2 days a week for 12 weeks for a 45 minute live, interactive strength training workout.
  Interventions: Behavioral: Vivo workout

INTERVENTIONS:
Behavioral: Vivo workout — 2 days a week for 12 weeks of a live, interactive virtual strength training program. Each class is 45 minutes long and lead by a certified trainer.

SUMMARY:
This research trial studies the effect of an online, live and interactive strength training program on physical function and strength in older adults with prediabetes.

DETAILED DESCRIPTION:
It is well established that in-person resistance training is an effective form of exercise to increase physical function and quality of life amongst adults. However, older adults report not participating in resistance training due to lack of age appropriate programs, fear of a gym setting, poor access to a gym, joint and other kinds of pain, and lack of social support. These barriers have been compounded as a result of COVID-19 pandemic, wherein older adults are encouraged to socially isolate, leading to even less physical activity. Vivo is a virtual small group exercise program designed for adults 55 and addresses these major barriers to strength training by coaching through an interactive online training session incorporating social support and social engagement.

The investigators plan is to test a highly attractive technology platform specifically designed to meet the needs of older adults to demonstrate that resistance training exercise can be scaled and effective with diverse older adults and remove the barrier of having to go to a gym setting to see benefits. The investigators will test feasibility in a real world sample of adults ≥60 with prediabetes, a very prevalent, serious and often silent health condition that affects 1 in 3 adults in the US and is associated with high rates of sarcopenia, or loss of muscle mass.

In the next study, Phase II NCT06458530, investigators will examine the effects of Vivo on physical function and glycemic level in sedentary older with prediabetes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;

  * Diagnosis of Pre-diabetes within prior 12 months: fasting glucose between 100 to 126 OR HbA1c between 5.7 and 6.4%
  * Ambulatory and community-dwelling
  * Sedentary: less than 150 minutes of moderate physical activity OR less than 75 minutes of vigorous physical activity per week
  * Have not engaged in resistance training for at least 6 months prior to enrollment
  * Low functioning (defined as able to do at least 1 chair stand without using hand in 30 second but unable to meet the moderate function criteria for age and gender)
  * Access to WiFi (or internet connection) in defined exercise space
  * Willing to maintain weight and current diet throughout the study

Exclusion Criteria:

* Inability to complete physical function assessment or inability to do a chair stand without using hands.
* Use of antidiabetic medications
* Use of testosterone supplement or replacement
* Clinical disorder precluding/interfering with participation or assessments

  * Unstable angina, arrhythmia, uncontrolled hypertension
  * End Stage Renal Disease on Hemodialysis
  * Lower extremity amputation or paralysis
  * Neurological conditions causing functional or pronounced cognitive impairments
  * Active malignancy except for non-melanomatous skin cancers
* Unable to provide consent
* Weight instability

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from electronic medical records in Duke Maestro Care as described in the Clinical Trials Information. All participants who enrolled and were eligible for the trial participated in the feasibility study.
Groups:
- Vivo Intervention: Participants participated via Zoom in a virtual exercise class 2 days/week for 45 minutes for 12 weeks. Exercise classes were led by a certified trainer and each class focused on building strength, flexibility, balance, and cognitive skills
Period: Overall Study
Arm/Group | Vivo Intervention
Started | 28
Completed | 22
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Leg strength assessed through a 30 second chair rise test [Mean (Standard Deviation); unit: chair stands] | 12.1 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Leg Strength Assessed Through a 30 Second Chair Rise Test
Description: Participants completed as many chair stands as they could in 30 seconds
Time Frame: at 3 months (endpoint)
Measure: Mean (Standard Deviation); unit: number of chair stands
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
number of chair stands | 14.2 (2.9)

2. Primary Outcome: Workout Attendance
Description: Attendance to each workout session was tallied. A possible 24 workout sessions were offered for the intervention (12 weeks of 2 days a week for workouts). The number of participants includes everyone who completed intervention, excluding those who stopped intervention at some point. The data reported represents the overall percent attendance of the participants that completed the intervention (N=22 participants). Attendance was calculated by averaging the number of sessions attended divided by the total number of exercise sessions attended (24 sessions).
Time Frame: after each workout session for up to 3 months (endpoint)
Population: 22 participants completed the intervention. Each participant had the opportunity to attend 24 exercise sessions. The attendance rate was calculated based on the number of sessions the participant attended divided by the total possible sessions (24 sessions). The attendance rate was then averaged across the participants who completed the intervention.
Measure: Mean (Full Range); unit: percent of attendance
Units Other Than Participants: exercise sessions
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
Number analyzed (exercise sessions) | 24
percent of attendance | 85 [0 to 100]

3. Primary Outcome: Intervention Engagement Assessed by Self- Reported Ease of Use
Description: Participants completed a questionnaire (Likert Scale) on their experience using Vivo. 1= Strong Disagree to 5= Strongly Agree
Time Frame: at 3 months (endpoint)
Measure: Number; unit: percent of participants
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
percent of participants
  Easy to sign into class | 82
  Easy to follow workout instructions during class | 86
  Level system made it easy to tailor intensity and exercises to my abilities | 95

4. Primary Outcome: Program Satisfaction
Description: Participants completed the question on a questionnaire to answer "What was your overall satisfaction with Vivo?" Responses are percentage of participant who reported being satisfied or very satisfied with the Vivo intervention. A higher number indicates higher satisfaction.
Time Frame: at the 3 month (endpoint)
Measure: Number; unit: percent of participants
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
percent of participants | 95

5. Primary Outcome: Exercise Intervention Trainer Fidelity Checklist
Description: The exercise intervention fidelity as assessed at 4 time points over the course of the 12-week exercise program using a 9-item checklist to ensure unbiased assessment. The purpose was to observe the exercise session to see if the main areas of the intervention were being delivered; workout intensity, safety, and participation and engagement. The results below indicate the percentage of exercise workouts that met the 9-item checklist. A higher score indicates higher fidelity.
Time Frame: over the course of the 12 week intervention
Population: There were 4 exercise cohorts in this feasibility study, taught by different trainers. To ensure exercise fidelity across the cohorts, 4 exercise sessions from each cohort were observed for a total of 16 observed exercise sessions. A 9-item checklist was used to ensure components of the sessions were being met. The 16 sessions met 96% of the checklist components.
Measure: Number; unit: percentage of workouts meeting checklist
Units Other Than Participants: exercise sessions
Arm/Group | Vivo Strength Training
Number analyzed (Participants) | 22
Number analyzed (exercise sessions) | 16
percentage of workouts meeting checklist | 96

6. Other Pre Specified Outcome: Health-related Quality of Life Measured Via the Short Form (SF)-36
Description: Change from baseline to 3 months will be assessed (scores range from 0-100 with higher scores indicating better health-related quality of life)
Time Frame: baseline and at 3 months (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-12

7. Other Pre Specified Outcome: Satisfaction With Life Measured by the 5 Item SWL Questionnaire
Description: Changes from baseline to 3 months (SWL scores range from 5-35 with higher score indicating greater SWL)
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2025-12

8. Other Pre Specified Outcome: Profile of Mood Survey (POMS)
Description: Changes from baseline to 3 months will assess participant's changes in mood.
Time Frame: baseline and at 3 months (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-12

9. Other Pre Specified Outcome: Perceived Stress Scale Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Changes from baseline to 3 months will assess participant's changes in perceived stress. likert scale from 0-4, higher scores indicate higher stress
Time Frame: baseline and at 3 months (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-12

10. Other Pre Specified Outcome: Exercise Efficacy
Description: Changes from baseline to 3 months will be assessed using a questionnaire measuring the participant's confidence in completing exercise related behaviors
Time Frame: baseline and at 3 months (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-12

11. Other Pre Specified Outcome: Sleep Measured Via the Pittsburgh Sleep Quality Index (PSQI)
Description: Change from baseline to 3 months (PSQI scores range from 0-21 with higher scores indicating worse sleep quality)
Time Frame: baseline and at 3 months (endpoint)
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from enrollment to study completion or study withdraw. The duration of participation in the study was approximately 12 weeks.
Arm/Group | Vivo Intervention
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivo Intervention (N=22)
COVID infection (Infections and infestations) | 1 (1)
Back pain following a skiing accident (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain following exercise (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT05497960/Prot_SAP_000.pdf